CLINICAL TRIAL: NCT06699654
Title: Comparative Study Between Spirulina Gel and Spirulina Nanoparticles Gel for Treatment of Stage II Grade B Periodontitis: Randomized Control Clinical Study with Radiological and Biochemical Assessment
Brief Title: "Comparison of Spirulina Gels for Treating Stage II Grade B Periodontitis"
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Samir Mohamed Ahmed Algarf, B.D.S. (2017) Misr University for Science and Technology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-68
Record Dates: First submitted 2024-11-16; First posted 2024-11-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis Stage II
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three arms: Spirulina Gel, Spirulina Nanoparticles Gel, or control. The interventions are administered over a defined period with radiological and biochemical assessments conducted at baseline and post-treatment.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (control group) (Placebo Comparator): Participants in this arm will receive oral hygiene instruction and full mouth SRP of all teeth plus placebo gel instillation in the pocket.
  Interventions: Other: Placebo gel
- Group II (experimental I) (Active Comparator): Participants in this arm will receive oral hygiene instruction and full mouth SRP of all teeth followed by insertion of the spirulina gel instillation in the deepest selected periodontal pocket after drying the area around it.
  Interventions: Dietary Supplement: Spirulina Gel
- Group III (experimental II) (Experimental): Participants in this arm will receive oral hygiene instruction and full mouth SRP of all teeth followed by insertion of the spirulina nanogel instillation in the deepest selected periodontal pocket after drying the area around it.
  Interventions: Dietary Supplement: Spirulina Nanoparticles Gel

INTERVENTIONS:
Other: Placebo gel — A gel without active Spirulina components applied as a control intervention.
  Arms: Group I (control group)
Dietary Supplement: Spirulina Gel — A conventional Spirulina gel formulation applied as a periodontal therapy.
  Arms: Group II (experimental I)
Dietary Supplement: Spirulina Nanoparticles Gel — A novel Spirulina nanoparticles gel formulation applied as a periodontal therapy.
  Arms: Group III (experimental II)

SUMMARY:
This randomized controlled clinical study investigates the effectiveness of Spirulina gel and Spirulina nanoparticles gel in treating Stage II Grade B periodontitis. The research aims to compare the two formulations in terms of clinical, radiological, and biochemical outcomes, such as pocket depth reduction, alveolar bone density improvement, and inflammatory marker levels. The study seeks to provide insights into the potential of Spirulina-based therapies for enhancing periodontal health.

ELIGIBILITY:
Inclusion criteria:

* Patients with good systemic health.
* Patients who can maintain good oral hygiene.
* Attachment loss 3-4 mm and probing pocket depth ≤ 5mm. Exclusion criteria for this study include: ·

  * Any systemic disease that affects the periodontium. ·
  * Pregnant, postmenopausal women. ·
  * People who take anti-inflammatory drugs, antibiotics, or vitamins within the previous 3 month.
  * People who use mouth washes regularly ·
  * Participation in other clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Probing Pocket Depth (PPD) | at baseline, 1 month , 3 months, 6 months
  The mean reduction in probing pocket depth in millimeters (mm) at periodontal sites treated with Spirulina gel and Spirulina nanoparticles gel.

SECONDARY OUTCOMES:
Radiographic Bone Density Improvement | at baseline and after 6 months
  Changes in alveolar bone density measured using radiographic imaging techniques.
Biochemical Marker Levels | Measured at baseline, 1 month ,3 months, and 6 months
  Reduction in inflammatory markers specifically Superoxide dismutase enzyme levels in gingival crevicular fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Elgendy, Prof.Dr, Study Director — Kafrelsheikh University
Locations (1):
- Doctor Mohamed Samir Periodontal and Implantology Clinic, El-Sheikh Zayed City, Cairo Governorate, Egypt